CLINICAL TRIAL: NCT02501681
Title: Evaluation of Different Priming Solutions Effects on Microcirculation, Oxidative Stress and Morbidity in Cardiovascular Surgery Patients
Acronym: Acibadem
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Matty Koopmans, MSc, Frisius Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Atadek 2014-723
Record Dates: First submitted 2015-07-13; First posted 2015-07-17 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Microcirculation
Keywords: sublingual microcirculation; cardiovascular surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- crystalloid (Active Comparator): Group A (n=20); crystalloid as priming solution used in patients,
  Interventions: Other: priming solution during cardiovascular surgery
- colloid (Active Comparator): Group B (n=20); colloids as priming solution used in patients
  Interventions: Other: priming solution during cardiovascular surgery

INTERVENTIONS:
Other: priming solution during cardiovascular surgery

SUMMARY:
Single-centre prospective randomized study will be included the patients who undergo elective cardiovascular surgery. Preoperative fluid deficit will be calculated by the formula as starvation period X 4 X weight. Patients will be divided into two groups: Group A (n=20); crystalloid as priming solution used in patients, Group B (n=20); colloids as priming solution used in patients. In addition to priming solutions, extracorporeal pump will be filled with 150 mL of Mannitol, 60 mL of NaHCO3 and 10000 IU Insulin. Standard anesthesia protocol will be administered to all patients. Ringer's Lactate will be given at first 30 minute after induction. Ringer's Lactate as fluid maintenance will be administered at a rate of 100 mL/h except in extracorporeal circulation. Goal-directed fluid management will be performed by PVI (Pleth Variability Index). Cut off level of PVI will be accepted %15.

DETAILED DESCRIPTION:
For integrative investigation of the effects of priming solution and postoperative fluid management on the complex interrelation between microcirculation and reactive oxygen species; sublingual microcirculation using microcirculation imaging system (IDF, Cytocam, NL) will be displayed and measure ekstra vascular lung water (EVLW) using PiCCO and plasma levels of oxidative stress markers will be measured. Sublingual tissue microcirculation will be evaluated in all patients at different time points as before induction (T0), after induction (T1), before cross clamping-hypothermic period (T2), after cross clamping (T3), before end of pump (normothermic period, heating) (T4), acceptance to intensive care unit (T5), third hour after surgery (T6) and twenty forth hour after surgery (T7).

ELIGIBILITY:
Inclusion Criteria:

* cardiovascular surgery needed

Exclusion Criteria:

* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
change in microvascular flow index (MFI) | 1 day
  hemodilution by the priming solutions in extracorporeal circulation affects the sublingual microcirculation

SECONDARY OUTCOMES:
difference in MFI | 1 day
  differences can be detected in the microcirculatory response to crystaloid priming in relation to colloid (starch) priming.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Centre Leeuwarden, Leeuwarden, Netherlands